CLINICAL TRIAL: NCT03183167
Title: Universitätsklinikum Erlangen Cohort of Patients With Spontaneous Intracerebral Hemorrhage
Brief Title: Longitudinal Cohort Study on ICH Care
Acronym: UKER-ICH
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: Longitudinal study ICH care
Record Dates: First submitted 2017-06-06; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Spontaneous Intracerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
Intracerebral hemorrhage [ICH] is the most feared sub-type of stroke, associated with a high mortality rate up to 50% and thus leaving large proportions of patients in functionally dependent states. In recent years randomized trials have failed to provide an effective intervention to improve functional outcome in ICH. Therefore, evidence regarding acute therapeutic interventions as well as secondary treatment approaches is still limited.

The present monocentric longitudinal study on spontaneous ICH patients is based on a prospective institutional stroke registry including all hemorrhagic stroke patients treated at a German University Hospital, Department of Neurology, over a 10 year time frame (2006-2015). The main aim of this investigation, besides analyses of epidemiological aspects, will be (i) to identify possible treatment targets influencing functional outcome, and (ii) to evaluate existing therapeutic strategies in ICH care.

DETAILED DESCRIPTION:
Stroke is one of the leading causes for death and disability in the industrialized world. Intracerebral hemorrhage [ICH] represents one sub-type with a rather poor prognosis. As randomized trials of recent years failed to establish an effective treatment strategy in ICH, identification of therapeutic strategies is urgently needed. Furthermore, evidence on commonly carried out management approaches is limited and remains to be specifically established. Roughly, one third of patients experience hematoma enlargement strongly impacting functional outcome, yet hemostatic treatments have not shown to be safe and aggressive blood pressure reductions are safe but not significantly effective. Therefore, improved risk-stratification for patients at high-risk for hematoma growth may increase the effect size of possible interventions. Intraventricular hemorrhage initially present or occurring during hematoma growth may represent another therapeutic target as a potentially treatable outcome predictor, recently studied in the CLEAR-IVH trial. Again, functional outcome was not improved in favour of the intervention emphasizing the need to identify patients who may benefit the most. Furthermore, several management issues remain to be elucidated in critically ill ICH patients, i.e. how to prevent venous thrombosis or systemic thromboembolism, what is the impact of invasive intracranial pressure monitoring, how to prevent or treat peri-hemorrhagic edema and what is the role of surgical approaches?

This observational cohort study will try to strengthen the therapeutic evidence for ICH treatment by generating a large (n>1000) cohort of consecutive ICH patients treated a tertiary care hospital in Germany. Further, collaborative efforts will be undertaken to integrate and compare data from the present study to existing cohorts to validate specific findings. Patients will be identified from an institutional prospective stroke registry by the diagnosis of spontaneous primary ICH during a time period from 2006-2015. Only patients with spontaneous primary ICH will be included, other secondary etiologies will be excluded: i.e. tumors, trauma, vascular malformations, anticoagulation at presentation etc. will be excluded. Clinical data on demographics, medical history, pre-ICH medication exposures and laboratory results will be obtained by medical charts, institutional databases or prospective registries, supplemented by structured interviews or by review of all available medical records. Patient-derived follow-up information will be corroborated by review of pertinent medical records. An estimated total number of greater 1000 patients will be reviewed for this investigation. In detail the following parameters will be evaluated: - prior medical history (including CHADS-VASC-Score, HAS-Bled Score, vascular risk factors), - functional status prior admission (mRS), - neurological admission status (NIHSS, GCS), - imaging characteristics, - time intervals: symptom onset until admission, imaging, therapy initiation, - acute blood pressure management, - complications (hemorrhagic- or ischemic-events, infectious) and treatment (surgical treatment, mode of antithrombotic treatment or prophylaxis of systemic thromboembolism, intraventricular fibrinolysis, etc.), - mortality rates, - functional outcome (mRS);

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous Primary Intracerebral Hemorrhage

Exclusion Criteria:

* Secondary ICH etiology (i.e. AVM, SAH, SVT, Fistulas, Tumor, Trauma)
* ICH patients on active anticoagulation (known NOAC intake, INR Level on Admission >1.4)
* Patients with intraparenchymal hemorrhage after Thrombolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spontaneous Primary Intracerebral Hemorrhage
Sampling Method: Probability Sample
Enrollment: 1076 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Functional outcome | 90 days
  dichotomized by modified Rankin Scale 0-3 vs 4-6

SECONDARY OUTCOMES:
Hematoma enlargement | 24 hours
  ICH volume increase on Follow-up Imaging >33%
Intracranial complications | 90 days
  ischemic and hemorrhagic events
Extracranial complications | 90 days
  ischemic and hemorrhagic events
Functional outcome | 1 year
  dichotomized by modified Rankin Scale 0-3 vs 4-6

CONTACTS AND LOCATIONS:
Overall Officials: Hagen B. Huttner, MD. PhD., Principal Investigator — University Hospital Erlangen, Department of Neurology, Germany; Joji B. Kuramatsu, MD., Principal Investigator — University Hospital Erlangen, Department of Neurology, Germany
Locations (1):
- University or Erlangen-Nuremberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mrochen A, Song Y, Harders V, Sembill JA, Sprugel MI, Hock S, Lang S, Engelhorn T, Kallmunzer B, Volbers B, Kuramatsu JB. Influence of bundled care treatment on functional outcome in patients with intracerebral hemorrhage. Front Neurol. 2024 Aug 5;15:1357815. doi: 10.3389/fneur.2024.1357815. eCollection 2024. PMID 39161870
- [Derived] Sembill JA, Knott M, Xu M, Roeder SS, Hagen M, Sprugel MI, Mrochen A, Borutta M, Hoelter P, Engelhorn T, Rothhammer V, Macha K, Kuramatsu JB. Simplified Edinburgh CT Criteria for Identification of Lobar Intracerebral Hemorrhage Associated With Cerebral Amyloid Angiopathy. Neurology. 2022 May 17;98(20):e1997-e2004. doi: 10.1212/WNL.0000000000200261. Epub 2022 Mar 21. PMID 35314501
- [Derived] Sprugel MI, Kuramatsu JB, Volbers B, Saam JI, Sembill JA, Gerner ST, Balk S, Hamer HM, Lucking H, Holter P, Nolte CH, Scheitz JF, Rocco A, Endres M, Huttner HB. Impact of Statins on Hematoma, Edema, Seizures, Vascular Events, and Functional Recovery After Intracerebral Hemorrhage. Stroke. 2021 Mar;52(3):975-984. doi: 10.1161/STROKEAHA.120.029345. Epub 2021 Feb 1. PMID 33517701
- [Derived] Roeder SS, Sprugel MI, Sembill JA, Giede-Jeppe A, Macha K, Madzar D, Lucking H, Hoelter P, Gerner ST, Kuramatsu JB, Huttner HB. Influence of the Extent of Intraventricular Hemorrhage on Functional Outcome and Mortality in Intracerebral Hemorrhage. Cerebrovasc Dis. 2019;47(5-6):245-252. doi: 10.1159/000501027. Epub 2019 Jun 18. PMID 31212293